CLINICAL TRIAL: NCT04976842
Title: Acute Postoperative Pain in Opioid-free Anesthesia After Urological Procedures
Brief Title: Opioid-free Anesthesia and Acute Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Associate Professor of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OFA 1
Record Dates: First submitted 2021-07-10; First posted 2021-07-26 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia; Postoperative Pain; Cognitive Impairment, Variable
Keywords: ANESTHESIA; OPIOIDS; PAIN; COGNITIVE
MeSH Terms: conditions — Pain, Postoperative; Cognitive Dysfunction; Pain

STUDY DESIGN:
Intervention Model Description: 2 groups of patients assigned to either opioid-free anesthesia or opioid-based anesthesia were studied in a randomized manner as for postoperative pain and cognitive dysfunction
Who Masked: Participant, Outcomes Assessor
Masking Description: the investigator assessing outcome did not know the kind of anesthesia the patient received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-free anesthesia (Active Comparator): Opioid free anesthesia protocol for urological procedurs
  Interventions: Device: OFA
- Opioid-based anesthesia (Active Comparator): Opioid based anesthesia protocol for urological procedures
  Interventions: Drug: OBA

INTERVENTIONS:
Device: OFA — Anesthesiology technique based on Mulier protocol. Before induction, loading dose of dexmedetomidine 0,25mcg/kg (max 20mcg). Induction with dexmedetomidine 0,1mcg/kg, lidocaine 1mg/kg, ketamine 0,1mg/kg plus propofol 2mg/kg plus rocuronium1mg/kg IBW (if required). Maintenance with dexmedetomidine 0,1mcg/kg/h, lidocaine 1mg/kg/h, ketamine 0,1mg/kg/h and propofol infusion adjusted according to bispectral index indication ( BIS maintained 40-60). 15 minutes prior to end of surgery, the dose of drugs is reduced to dexmedetomidine 0,05mcg/kg/h, lidocaine 0,5mg/kg/h, ketamine 0,05mg/kg/h.
  Arms: Opioid-free anesthesia
Drug: OBA — Total intravenous anesthesia with propofol for maintenance of anesthesia. Fentanyl 2mcg/kg only at induction and infusion of propofol and remifentanil for maintenance, with doses adjusted according to bispectral index indication ( BIS maintained 40-60).
  Arms: Opioid-based anesthesia

SUMMARY:
Control of intraoperative and postoperative pain with the use of opioids constitutes normal practice. Opioid free anesthesia (OFA) is a relatively recent anesthesiology practice according to which opioids are not administered during surgery and are avoided postoperatively. Opioid free anesthesia seems to provide better quality of postoperative analgesia while protecting the patient from the side effects of opioids such as respiratory depression, postoperative nausea and vomiting (PONV), opioid induced hyperalgesia and postoperative cognitive dysfunction. The aim of this study is to investigate the possible difference in the intensity of postoperative pain (based on the numeric rating scale 0-10) and the presence of PONV in patients undergoing transurethral urologic surgery under general anesthesia, when patients receive randomly either opioid free anesthesia (OFA) or opioid based anesthesia (OBA).

DETAILED DESCRIPTION:
This study aimed to study postoperative pain after opioid free anesthesia or opioid based anesthesia after urologica; procedures. The two study groups opioid free (OFA) and opioid based (OBA) were as follows:

OFA: Anesthesiology technique based on Mulier protocol. Before induction, loading dose of dexmedetomidine 0,25mcg/kg (max 20mcg). Induction with dexmedetomidine 0,1mcg/kg, lidocaine 1mg/kg, ketamine 0,1mg/kg plus propofol 2mg/kg plus rocuronium1mg/kg IBW (if required). Maintenance with dexmedetomidine 0,1mcg/kg/h, lidocaine 1mg/kg/h, ketamine 0,1mg/kg/h and propofol infusion adjusted according to bispectral index indication ( BIS maintained 40-60). 15 minutes prior to end of surgery, the dose of drugs is reduced to dexmedetomidine 0,05mcg/kg/h, lidocaine 0,5mg/kg/h, ketamine 0,05mg/kg/h.

OBA: Total intravenous anesthesia with propofol for maintenance of anesthesia. Fentanyl 2mcg/kg only at induction and infusion of propofol and remifentanil for maintenance, with doses adjusted according to bispectral index indication ( BIS maintained 40-60).

Both groups receive ranitidine 50mg, dexamethasone 4 mg and paracetamol 1g iv 15 min before the end of surgery. Postoperative analgesia for both groups consists of paracetamol 3g/24h iv, rescue analgesia with tramadol 1mg/kg iv max x3, rescue for PONV ondacetron 4 mg iv.

The outcomes assessed were:

Primary outcome:

1. Intensity of acute postoperative pain (NRS 0-10), time frame up to 24h postoperatively
2. Nausea and vomiting

Secondary outcome:

1. Change in minimental state evaluation test, time frame pre-op, 1h post-op, at discharge
2. Severe postoperative adverse effect related to anesthesia (postoperative hypoxemia, ileus, postoperative cognitive dysfunction)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged>18 years old
* ASA I-III
* Patients scheduled for elective transurethral urologic surgery with general anesthesia

Exclusion Criteria:

* • Patient refusal

  * Use of opioids pre-op
  * Inability to read or write
  * Known psychiatric disease under medication
  * Dementia
  * Severe liver and renal disease
  * Known allergy to drugs used
  * Known arrhythmia (2nd-3rd AV block, acute unstable angina, acute myocardial infarction in the past 6 weeks or severe cardiac problem-condition)
  * Heart rate<45 bpm
  * Pre-op minimental test<23
  * Major surgery complications (hemorrhage with need for transfusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | baseline and 24 hours
  Intensity of acute postoperative pain (measured by numeric rating scale NRS 0-10), time frame up to 24h postoperatively

SECONDARY OUTCOMES:
postoperative cognitive dysfunction | baseline and 24 hours
  Change in minimental state evaluation test up to 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece